CLINICAL TRIAL: NCT01363102
Title: Effects of a Systematic Team Approach to Guide Early Mobilization in Surgical ICU Patients
Brief Title: Systematic Team Approach to Guide Early Mobilization in Surgical Intensive Care Unit Patients
Acronym: mSOMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of Massachusetts, Worcester (Other); Technical University of Munich (Other); University of Salzburg (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Director of Research, Surgical Intensive Care Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11112010
Record Dates: First submitted 2011-05-23; First posted 2011-06-01 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Muscle Weakness; Critical Illness; Respiratory Insufficiency
Keywords: Muscle strength; functional mobility; outcome; intensive care unit; quality of life
MeSH Terms: conditions — Muscle Weakness; Critical Illness; Respiratory Insufficiency | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Group will undergo usual mobilization per standard SICU care
- Study Group (Experimental): Patient mobilization discussed on rounds, SOMS score goal created, specific attempt to mobilize patient and achieve goal throughout day.
  Interventions: Procedure: SOMS

INTERVENTIONS:
Procedure: SOMS — Apply a number to mobilization goal for patient
  Other Names: Early Mobilization
  Arms: Study Group

SUMMARY:
The investigators hypothesize that by applying a validated algorithm to accomplish early mobilization in surgical intensive care unit (ICU) patients, these patients will achieve a higher level of mobility which translates to shorter ICU length of stay and improved functional status at discharge. Additionally, the investigators hypothesize that genetic polymorphisms related to muscle strength and sleep will also explain some variance in these outcome variables.

DETAILED DESCRIPTION:
The trauma literature consistently shows that early mobilization improves patients' outcome after a localized trauma such as hip fracture, or blunt solid organ injuries. In addition, in critically ill patients on the medical ICU, early mobilization improves patients' functional outcome and decreases ICU length of stay (1). This study evaluates if critically ill patients in a surgical ICU can safely and effectively be mobilized early after trauma and surgery. The investigators propose to conduct a randomized controlled study in surgical intensive care unit patients to evaluate the effects of mSOMS guided early mobilization. Additionally, the study will examine known genetic polymorphisms as related to sleep quality and muscle strength and how it relates to early mobilization of surgical ICU patients. In particular, the study will focus on the following polymorphisms: CLOCK, NPAS2, PER2 and PER3, PDE4D,MUC1, ATP2B1, DCDC5, TRPM6, SHROOM3, and MDS1 genes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or greater)
* Who have been on mechanical ventilation for less than 48 hours and are expected to continue for at least 24 more hours
* Who meet criteria for baseline functional independence (Barthel Index greater than or equal to 70 obtained from a proxy describing patient function 2 weeks before admission

Exclusion Criteria:

* Irreversible disorders with 6-month mortality greater than 50%
* Rapidly developing neuromuscular disease
* Cardiopulmonary arrest
* Motor component of Glascow Coma Scale <5
* Elevated intracranial pressure
* Ruptured/leaking aortic aneurysm
* Acute MI before peak troponin has been reached
* Absent lower limbs
* Pregnancy
* Unstable fractures contributing to likely immobility
* Hospitalization prior to ICU admission >5 days
* Enrollment in another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Average achieved SOMS level | Average SOMS level from time to inclusion to ICU discharge readiness, an expected time of one to two weeks (expected time of one to two weeks).
  Achieved SOMS level will be assessed daily and average values be taken for comparison between groups.

SECONDARY OUTCOMES:
SICU length of stay | Patients will be followed until SICU discharge, an expected 2 days to 2 weeks
  Time from study inclusion to SICU discharge readiness, an expected time of one to two weeks.
The "mini" modified Functional Independence Measure (mmFIM) level | mmFIM will be measured twice, at ICU discharge readiness and hospital discharge readiness, an expected average of one to two and three weeks, respectively.
  Using the modified Functional Independence Measure (mmFIM), the levels of the locomotion and transfer mobility domain at hospital discharge (4 point NRS) will be compared between groups.
Quality of life following hospital discharge | three months after hospital discharge
  SF 36 score
Muscle strength | ICU and hospital discharge readiness, an expected time of one to two and three weeks, respectively.
  Medical Research Council (MRC) scale.
Side effects of mobilization therapy | during and 30 minutes after mobilization therapy during SICU stay, approximately 1 to 2 weeks.
  Number of unfavorable signs and symptoms or unintended deterioration of clinical status associated with mobilization therapy, including, but not limited to, unplanned extubation or dislodgment of drains, arterial catheters, venous devices, or other medical equipment. The relationship of any untoward event to mobilization therapy was assessed by the clinician and reported as unrelated, unlikely, possibly, or definitely related. AE were also categorized by intensity as mild, moderate, or severe
Genetic Polymorphisms as related to the other outcomes | 5 minutes to collect sample
  Since Sleep duration has a genetic component corresponding to 40% heritability, we are going to conduct an analysis of known polymorphisms that are related to different variables of sleep quality and how it relates to muscle strength and mobility. In particular we will focus on polymorphisms in CLOCK, NPAS2, PER2 and PER3, PDE4D,MUC1, ATP2B1, DCDC5, TRPM6, SHROOM3, and MDS1 genes, which are associated with sleepiness, sleep phase, inertia, and potentially with respiratory muscle weakness and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — The Massachusetts General Hospital
Locations (5):
- United States (3):
  - The Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
- University of Salzburg, Salzburg, Austria
- Technische Universität München, München, Bavaria, Germany

REFERENCES:
- [Background] Kasotakis G, Schmidt U, Perry D, Grosse-Sundrup M, Benjamin J, Ryan C, Tully S, Hirschberg R, Waak K, Velmahos G, Bittner EA, Zafonte R, Cobb JP, Eikermann M. The surgical intensive care unit optimal mobility score predicts mortality and length of stay. Crit Care Med. 2012 Apr;40(4):1122-8. doi: 10.1097/CCM.0b013e3182376e6d. PMID 22067629
- [Derived] Schaller SJ, Anstey M, Blobner M, Edrich T, Grabitz SD, Gradwohl-Matis I, Heim M, Houle T, Kurth T, Latronico N, Lee J, Meyer MJ, Peponis T, Talmor D, Velmahos GC, Waak K, Walz JM, Zafonte R, Eikermann M; International Early SOMS-guided Mobilization Research Initiative. Early, goal-directed mobilisation in the surgical intensive care unit: a randomised controlled trial. Lancet. 2016 Oct 1;388(10052):1377-1388. doi: 10.1016/S0140-6736(16)31637-3. PMID 27707496
- [Derived] Meyer MJ, Stanislaus AB, Lee J, Waak K, Ryan C, Saxena R, Ball S, Schmidt U, Poon T, Piva S, Walz M, Talmor DS, Blobner M, Latronico N, Eikermann M. Surgical Intensive Care Unit Optimal Mobilisation Score (SOMS) trial: a protocol for an international, multicentre, randomised controlled trial focused on goal-directed early mobilisation of surgical ICU patients. BMJ Open. 2013 Aug 19;3(8):e003262. doi: 10.1136/bmjopen-2013-003262. PMID 23959756